CLINICAL TRIAL: NCT06473220
Title: Evaluation of the Effectiveness of Narrative Nursing in Patients With Alzheimer's Disease
Brief Title: Evaluation of the Effectiveness of Narrative Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fang Honglian, Principal Investigator, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 310638478
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease; Narrative; Depression, Anxiety
MeSH Terms: conditions — Alzheimer Disease; Narration; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference group (Other): The reference group carried out routine nursing, that is, the most appropriate intervention measures were properly formulated according to the actual condition degree and various levels of physical fitness of the patients, and the patients were urged to take drugs according to the doctor's advice every day. Nurses should conduct oral health promotion for patients; Administering medication and a daily healthy diet regimen; Patients with orientation and language communication disorders were given nursing care step by step. Continuous care for 2 months.
  Interventions: Behavioral: Narrative nursing
- Study group (Experimental): The research group cooperated with the implementation of narrative nursing. The detailed measures are as follows: ① Establish a narrative nursing special group. ② Narrative data collection. ③ Pay attention to the scientific evaluation of narrative content. ④ Edit the narrative reasonably. ⑤ Strengthen interview intervention. Continuous care for 2 months.
  Interventions: Behavioral: Narrative nursing

INTERVENTIONS:
Behavioral: Narrative nursing — Narrative nursing is an intervention mode of psychological nursing.

SUMMARY:
To explore the effects of narrative nursing on mental state, life ability and emotion of patients with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
There is no effective clinical treatment, mainly through taking Western drugs to control the Alzheimer's disease, but the treatment cycle is long, the cost of drugs is high, and the patient's family nee care, resulds long-termting in a huge economic and psychological burden on the patient and family recipients. Narrative nursing is an intervention mode of psychological nursing.In practice, narrative nursing can guide patients to actively organize experiences into various events with certain practical significance, attach importance to personal feelings and experiences, promote the psychological growth of patients and promote the generation of upward motivation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Alzheimer's Disease.
2. Forgetting is the main cognitive impairment;.
3. The patient has basic language communication ability.
4. Patients were treated with the same regimen.

Exclusion Criteria:

1. Patients with other common neurological and mental disorders (depression, psychosis, vascular cognitive impairment).
2. Patients with heart, liver and other vital organ dysfunction.
3. Patients with severe cardiovascular disease.
4. Patients with severe physical disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
MMSE sore | After 1, 2 and 4 weeks after hospitalization
  The simple mental state Intelligence Scale (MMSE) was used to evaluate the mental state of the patients before and after the nursing intervention. The scale was mainly composed of 5 dimensions, namely orientation ability, recall ability, memory ability, attention and calculation ability, and language ability, and contained a total of 30 items. The total score was 0-30 points, the higher the score, the better the mental state of the patients.
ESCA score | After 1, 2 and 4 weeks after hospitalization
  The self-care ability measurement (ESCA) scale was used to evaluate the practical self-care ability of patients in the two groups before and after nursing intervention. The scale was mainly composed of four dimensions: self-concept, health knowledge mastery level, sense of responsibility, and self-care practical skills, and contained 43 items with a total score of 0-172. It shows that the actual ability of self-care is better.
HAMD score | After 1, 2 and 4 weeks after hospitalization
  The score consisted of 17 items, including self-awareness, work and interest, gastrointestinal symptoms, weight loss, hypochondriasis, sleep difficulty, etc. The total score < 7 was considered normal, 7 to 17 divided into possible depression syndrome, > 17-24 were classified as having depression, and> 24 were classified as major depression.
HAMA score | After 1, 2 and 4 weeks after hospitalization
  The score includes two dimensions: spirituality and physicality, with a total of 14 items, including gastrointestinal and digestive symptoms, depressive mood, sensory system symptoms, behavioral manifestations when communicating with others, somatic anxiety, cognitive function, etc. The total score is > 28, which is classified as severe anxiety, 21 to 28 grades are anxious, 14 to < 21 is classified as anxiety, 7 to < 14 scores may have anxiety, and <7 is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Huang C ying, Bachelor, Study Chair — The Affiliated Brain Hospital of Nanjing Medical University
Locations (1):
- Gulou District, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Respect privacy rights.